CLINICAL TRIAL: NCT06395298
Title: Effects of the Application of PIOMI (Premature Oral Motor Intervention) in the Oral Feeding of the Premature: Randomized Clinical Trial
Brief Title: Effects of the Application of PIOMI in the Oral Feeding of Premature
Acronym: PIOMI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Sant Joan de Déu (Other)
Collaborators: Sociedad Espanola de Gastroenterologia, Hepatologia y Nutricion Pediatrica (Other); Nexe Foundation (Unknown); University Ramon Llull (Other); Borja Institute of Bioethics (Unknown); Institut de Recerca Sant Joan de Déu (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C.I.PIC-108-22
Record Dates: First submitted 2023-01-09; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Dysphagia; Disorder; Feeding, Newborn; Premature
Keywords: Swallowing; Swallowing disorders; Nutritional support; Feeding disorders; Preterm; Neonates; Sucking Behavior
MeSH Terms: conditions — Deglutition Disorders; Premature Birth; Feeding and Eating Disorders; Sucking Behavior

STUDY DESIGN:
Intervention Model Description: * Assignment: Random and parallel using the OxMaR (Oxford Minimization and Randomization) software
  * Age range: 29-30 gestational weeks, both sexes will participate
    * Control group:
  Will receive the traditional intervention model of the Neonatal Intensive Care Unit (non-nutritive suction and kangaroo method)
  o Experimental group: Application of the PIOMI (Premature Infant Oral Motor Intervention) protocol, for 5 minutes twice a day, in a period of 10 days o Both groups will receive gustatory and olfactory stimulation
  * Intervention model: Parallel assignment
  * Description of the intervention model: Comparison of two groups, treated with the application of the care model in the NICU (Neonatal Intensive Care Unit) and the application of PIOMI (Premature Infant Oral Motor Intervention)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: * Masking: Double blind
  * Masking methodology:
  The Sant Joan de Déu Hospital Neonatal Unit carries out its care activity under the NIDCAP model, which includes care centered on the user and the family/mother or caregiver.
  Currently, the design of the neonatal unit has individual boxes for the family member, which will allow the intervention to be carried out, as well as the orientations carried out by the health personnel with privacy and thus avoiding the identification of the different intervention models.
  For the realization of the blind, it is proposed to make two video capsules in which the activities to be carried out will be collected, both by the control group and the experimental group, interspersing in the case of the experimental the PIOMI activities with the basic nursing care without doing reference to the intervention model assigned in the recording. Access to the video will be in quick response code format.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group PIOMI (Experimental): Participants will receive:
  1. The traditional intervention Newborn Individualized Development Care and Assessment Program (NIDCAP) model of the Neonatal Intensive Care Unit (NICU) .The nurse providing direct care to the patient and family, will carry out the relevant care of the patient.
  2. The Premature Oral Motor Intervention (PIOMI) .The family will apply the PIOMI , 7 activities are intraoral stimulation for 10 consecutive days, twice a day, 5 minutes.
  3. Gustatory stimulation technique:the application of oropharyngeal colostrum, a 0.5 milliliter twice a day
  4. Olfactory stimulation Technique:A swab is moistened in breast milk and placed near the nose for one minute, twice a day.
  Interventions: Other: Experimental group PIOMI
- Control Group NIDCAP (Sham Comparator): Participants will receive :
  1.The traditional intervention Newborn Individualized Development Care and Assessment Program (NIDCAP) model of the Neonatal Intensive Care Unit (NICU).The nurse providing direct care to the patient and family, will carry out the relevant care of the patient.
  3.Gustatory stimulation technique:the application of oropharyngeal colostrum, a 0.5 milliliter twice a day
  4.Olfactory stimulation Technique:A swab is moistened in breast milk and placed near the nose for one minute, twice a day.
  Interventions: Other: Control group NIDCAP

INTERVENTIONS:
Other: Experimental group PIOMI — A group treated with the application of the care model Newborn Individualized Development Care and Assessment Program (NIDCAP) in the Neonatal Intensive Unit Care (NICU)+PIOMI
  Other Names: PIOMI+NIDCAP
  Arms: Experimental Group PIOMI
Other: Control group NIDCAP — A group treated with the application of the care model Newborn Individualized Development Care and Assessment Program (NIDCAP) in the Neonatal Intensive Unit Care (NICU)
  Other Names: NIDCAP
  Arms: Control Group NIDCAP

SUMMARY:
The goal of this clinical trial is assess whether the application of the premature oral motor intervention (PIOMI) combined with the Newborn Individualized Developmental Care and Assessment Program (NIDCAP), allows withdrawal of the external feeding device with guarantees of the patient's nutritional status, determining breastfeeding rates at hospital discharge and swallowing safety earlier than if only the care activity corresponding to the NIDCAP model is carried out, as well as the applicability of this standardised protocol in the neonatal intensive care unit of a tertiary hospital.

DETAILED DESCRIPTION:
Prematurity is one of the most common factors affecting the development of oromotor skills, interfering with feeding. The most common clinical manifestation is uncoordinated sucking-breathing-swallowing cycle.

The incidence of oropharyngeal dysphagia in paediatrics is estimated at 10.40%, doubling in preterm infants weighing less than 1500 grams. The aetiological distribution of swallowing disorders in the neonatal age is highly variable, as is their clinical presentation. Current literature reflects the impact of the use of an external feeding device on the quality of life of the patient-family, as well as the increased health care costs due to prolonged hospitalisation, emergencies for device removal, consumables and enteral nutrition.

Current health models are based on prevention, hence the importance of establishing early protocols for assessment, diagnosis and intervention. The main difficulty in neonatal intensive care units is the loss of opportunity for oral feeding and the absence of standardised protocols, as there is great controversy regarding the intervention techniques that should be applied to promote the development of oral-motor skills.The PIOMI is the intervention model that currently presents the greatest scientific production, the results obtained in the studies carried out show a high success rate in relation to the initiation of oral feeding in preterm infants, as well as the maintenance of high breastfeeding rates at the time of hospital discharge and at 10 days, in compliance with the standards of the World Health Organisation (WHO).

At present, there are study designs of PIOMI, combined with olfactory-gustatory stimulation, but the latter is not specified as an oropharyngeal colostrum technique, which is currently indicated in the therapeutic guidelines, nor is the protocolised nursing care model described, an aspect that is of great importance because each hospital centre offers different care depending on whether or not the model is based on the individualised assessment and care programme for the development of the newborn.

This research aims to evaluate these aspects by means of a randomised double-blind parallel allocation clinical trial using Oxford Minimization and Randomization (OxMaR) software, to be carried out at the Hospital Sant Joan de Déu in Barcelona, in the neonatal intensive care unit in the period November 2023-2026. The sample size is n=35 preterm infants of gestational age 29-30+6.

The control group will follow the NIDCAP care model and the experimental group will apply the PIOMI+NIDCAP protocol for 5 minutes twice a day for 10 days, with olfactory stimulation and oropharyngeal colostrum for both groups.

The family will apply the intervention by accessing a quick response code with an information capsule according to the assigned group.

To identify factors, sociodemographic and health variables, process variables and outcome variables will be selected using the Neonatal Oral-motor Assessment Scale (NOMAS), Early Feeding Skills Assessment (EFSA) and pre- and post-tests will be analysed using variance analysis program (ANOVA) and statistical package for the social sciences (SPSS)

ELIGIBILITY:
Inclusion Criteria:

* Neonates born at the Sant Joan de Déu Hospital with a gestational age between 29-30 weeks carrying an external feeding device due to the difficulty of oral feeding and that the medical team in charge considers clinically stable.

Exclusion Criteria:

* Endotracheal intubation or high-flow ventilatory support.
* Exclusive parenteral nutrition.
* Hyporeactive due to the use of sedative drugs.
* Condition of prematurity associated with other pathologies (syndromes, acquired brain damage, gastrointestinal malformations, airway and craniofacial malformations).

Ages: 29 Weeks to 30 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Estimated)
Dates: Start 2023-02-13 (Actual); Primary Completion 2026-06-03 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Time to remove the external feeding device | Days of life of the baby when the external feeding device is removed assessed up to 30 days
  To perform a proper calculation, the investigator must quantify the days of life in which the feeding device is placed and the date of effective removal

SECONDARY OUTCOMES:
Volume of intake at discharge | Milliliters that the baby take orally until the day of hospital discharge up to 4 weeks
  To perform a proper calculation, the investigator must quantify the volumen of milk in millilitres from the day of device removal until hospital discharge.
Hospitalization days | Days that the premature baby remains hospitalized from birth to hospital discharge up to 12 weeks
  Quantify the days from birth to hospital discharge.
Breastfeeding patients after hospital discharge | Number of patients who are breast-feeding after hospital discharge up to 12 weeks
  Quantify the babies who perform Breastfeeding, Deferred breastfeeding or Artificial Breastfeeding according to the group assigned at discharge.
Deferred breastfeeding patients after hospital discharge | Number of patients who are Deferred breast-feeding after hospital discharge ,up to 12 weeks
  Quantify the babies who perform Breastfeeding, Deferred breastfeeding or Artificial Breastfeeding according to the group assigned at discharge
Formula feeding patients after hospital discharge | Number of patients who are formula feeding after hospital discharge, up to 12 weeks
  Quantify the babies who perform Breastfeeding, Deferred breastfeeding or Artificial Breastfeeding according to the group assigned at discharge.
Weight at hospital discharge | Assess weight discharge day, up to 12 weeks
  To estimate the existence of significant differences between the group that presented intervention and the control.
Weight ten days at hospital discharge | Assess weight ten days at hospital discharge, up to 12 weeks
  Differences between discharge and 10-day weights

OTHER OUTCOMES:
Results of the items of the evaluation Neonatal Oral-Motor Assessment Scale (NOMAS) | The researchers will administer Neonatal Oral-Motor Assessment Scale (NOMAS)last day of intervention(10 days)
  The NOMAS tool consists of 29 items distributed in 3 domains:
  * Normal pattern: The range is from 27 to 40, with 27 being the lowest score and 40 being the highest score.
  * Disorganized pattern:The range is from 14 to 26, with 14 being the lowest score and 26 being the highest score.
  * Disfunctional pattern:The range is from 0 to 14, with 0 being the lowest score and 14 being the highest score.
  To achieve the feasibility of the evaluation tools Neonatal Oral-Motor Assessment Scale (NOMAS), the percentage of responses obtained will be taken into account. As a descriptive data analysis tool, the International Business Machines (IBM)software, Statistical Package for Social Sciences(SPSS) version 19.0.1 and variance analysis program(ANOVA), will be used in the pre- and post-test comparative data analysis.
Results of the items of the evaluation Early Feeding Skills (EFS) | The researchers will administer (EFS)last day of intervention (10 days)
  The EFSA tool consists of 19 items distributed in 5 domains:
  Regulation of breathing 5 items: The range is from 5 to 15 with 5 being the lowest score and 15 being the highest score
  Oromotor function 4 items: The range is from 4 to 12 with 4 being the lowest score and 14 being the highest score
  Swallowing-breathing coordination 4 items: The range is from 4 to 12 with 4 being the lowest score and 12 being the highest score
  Attention when taking 2 items and stability: The range is from 2 to 6 with 2 being the lowest score and 6 being the highest score
  Physiological 4 items: The range is from 4 to 12 with 4 being the lowest score and 12 being the highest score
  To achieve the feasibility of the evaluation tools EFS, the percentage of responses obtained will be considered. As a descriptive data analysis tool, Statistical package for the social sciences version 19.0.1 and variance analysis program, will be used in the pre- and post-test comparative data analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Raquel García Ezquerra, Principal Investigator — Sant Joan de Déu Hospital; Vanesa Ejarque Marin, Principal Investigator — Sant Joan de Déu Hospital
Locations (1):
- Raquel García Ezquerra, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Initially, the researchers plan to share the study protocol, the statistical analysis and the summary of results obtained, both in congresses and in publications, if applicable.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 1 year

REFERENCES:
- [Background] Grassi R, Farina R, Floriani I, Amodio F, Romano S. Assessment of fetal swallowing with gray-scale and color Doppler sonography. AJR Am J Roentgenol. 2005 Nov;185(5):1322-7. doi: 10.2214/AJR.04.1114. PMID 16247157
- [Background] Ghomi H, Yadegari F, Soleimani F, Knoll BL, Noroozi M, Mazouri A. The effects of premature infant oral motor intervention (PIOMI) on oral feeding of preterm infants: A randomized clinical trial. Int J Pediatr Otorhinolaryngol. 2019 May;120:202-209. doi: 10.1016/j.ijporl.2019.02.005. Epub 2019 Feb 5. PMID 30851536
- [Background] Lessen BS. Premature infant oral motor intervention (PIOMI) translating interventional research into interdisciplinary practice [Internet]. Unpublished; 2012. Disponible en: http://dx.doi.org/10.13140/RG.2.1.3652.696
- [Background] Shailaja S J, Jayashri S K. Comparative study on the effect of oral motor intervention protocols on oral motor skills of preterm infants from tertiary care hospital in metropolitan city: pilot study. Int J ContempPediatr [Internet]. 2020;7(7):1506.
- [Background] Tian X, Yi LJ, Zhang L, Zhou JG, Ma L, Ou YX, Shuai T, Zeng Z, Song GM. Oral Motor Intervention Improved the Oral Feeding in Preterm Infants: Evidence Based on a Meta-Analysis With Trial Sequential Analysis. Medicine (Baltimore). 2015 Aug;94(31):e1310. doi: 10.1097/MD.0000000000001310. PMID 26252313
- [Background] Pickler RH, Best A, Crosson D. The effect of feeding experience on clinical outcomes in preterm infants. J Perinatol. 2009 Feb;29(2):124-9. doi: 10.1038/jp.2008.140. Epub 2008 Oct 2. PMID 18830247
- [Background] Boiron M, Da Nobrega L, Roux S, Henrot A, Saliba E. Effects of oral stimulation and oral support on non-nutritive sucking and feeding performance in preterm infants. Dev Med Child Neurol. 2007 Jun;49(6):439-44. doi: 10.1111/j.1469-8749.2007.00439.x. PMID 17518930
- [Background] Lessen BS. Effect of Oral Stimulation on Feeding Progression in Preterm Infants. Adv Neonatal Care [Internet]. 2009 Aug [cited 2021 Feb 14];9(4):187. Available from: https://journals.lww.com/00149525-200908000-00021